CLINICAL TRIAL: NCT05370937
Title: Clınıcal Results of Evelator and Free Knot Methods In Medial Menıscus Posterior Root Tears
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, güneş sarıkaya, Principal investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 31.03.2022
Record Dates: First submitted 2022-04-11; First posted 2022-05-12 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Meniscus Tear; Meniscus Lesion
Keywords: medial meniscus posterior root tear; transtibial pullout system

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ELEVATOR (Active Comparator): After knotting the posterior root of the medial meniscus with a fiber rope, a tunnel will be opened for the rope to pass through the medial of the proximal crest of the tibia. Then, arthroscopically, the rope will be taken through the joint and passed through the tunnel, and the knot will be fixed to the tibia by using the endobutton elevator system
  Interventions: Procedure: ARTROSCOPİC SURGERY WITH ELEVATOR SYSTEM
- FREE KNOT (Active Comparator): The first stage of fixation is the same, and fixation to the tibia will be done with an endobutton by tying a free knot without using an elevator system.
  Interventions: Procedure: ARTROSCOPİC SURGERY WITHOUT ELEVATOR SYSTEM

INTERVENTIONS:
Procedure: ARTROSCOPİC SURGERY WITH ELEVATOR SYSTEM — TRANSTİBİAL PULL OUT REPAİR FOR MEDİAL MENİSCUS POSTERİOR ROOT TEARS
  Arms: ELEVATOR
Procedure: ARTROSCOPİC SURGERY WITHOUT ELEVATOR SYSTEM — TRANSTİBİAL PULL OUT REPAİR FOR MEDİAL MENİSCUS POSTERİOR ROOT TEARS WITH ELEVATOR SYSTEM
  Arms: FREE KNOT

SUMMARY:
In this thesis study, the transtibial pullout method, which is one of the treatment methods for medial meniscus posterior root tear, will be used in patients over the age of 18 with medial meniscus posterior root tear, who applied to the Atatürk University Orthopedics and Traumatology clinic. The patients will be divided into two groups. In the first group, after knotting the posterior root of the medial meniscus with a fiber rope, a tunnel will be opened for the rope to pass through the medial of the proximal crest of the tibia. Then, arthroscopically, the rope will be taken through the joint and passed through the tunnel, and the knot will be fixed to the tibia by using the endobutton elevator system. In the second group, the first stage of fixation is the same, and fixation to the tibia will be done with an endobutton by tying a free knot without using an elevator system. The clinical and radiological scores of both groups just before the operation and at the twelve months after the operation will be calculated and their relationship with each other will be examined.

DETAILED DESCRIPTION:
This thesis study is planned as a prospective study and approximately 30 patients with medial meniscus posterior root tear over the age of 18 who will apply to Erzurum Atatürk University Research Hospital Orthopedics and Traumatology clinic are planned to participate in this study. Based on a study by Yuki et al. (reference 3), the difference in the Lysholm score in the first group, which will be fixed with the elevator system, in the preoperative and postoperative sixth month was 33± 10 units, and in the second group, the difference in the preoperative and postoperative sixth month was 20± 14 units to be statistically significant, it was calculated with the G*POWER 3.1.9.4 program that 15 patients from each group should be taken at 80% power and 95% confidence level, a total of 30 patients. Patients will be divided into two groups of 15 people each. The endobutton elevator system will be used in the tibial fixation of the first group. In the tibial fixation of the second group, the endobutton free knot technique will be used. Demographic information of the patients will be recorded. Vas score, Lysholm score and Kellgren-lawrance classification will be made for the patients in these two groups, according to the results of the outpatient clinic control just before the operation and at the twelve months after the operation. This will be done by a physician who is in our entire follow-up clinic and does not go into the surgery of the patients. The clinical scores and radiological degenerative changes of these two groups just before the operation and at the twelve months after the operation will be examined

ELIGIBILITY:
Inclusion Criteria:

1. older than 18 years
2. Findings showing medial meniscus root repair indication in the MRI with Outer-Bridge grade 1 or 2 and Kellegren Lawrence grade 0-2

Exclusion Criteria:

1. Patients with chronic knee pain and chronic use of NSAIDs or opioids
2. Patients with chronic instability and anterior cruciate ligament damage in addition to medial meniscus root tear
3. Patients who had meniscus root repair before, but did not get good results and went for revision
4. Patients who underwent tibial osteotomy with meniscus root repair.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-10-16 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-04-16 (Actual)

PRIMARY OUTCOMES:
Lysholm score | immediately before the surgery to 12-month post-operative period
  0-100-The Lysholm score is a 100-point scoring system for examining a patient's knee-specific symptoms including mechanical locking, instability, pain, swelling, stair climbing, and squatting.
Visual analoque score | immediately before the surgery to 12-month post-operative period
  (0-10, 0=no pain, 10=worst imaginable pain)
Tegner Activity Score | immediately before the surgery to 12-month post-operative period
  The Tegner activity scale is a one-item score that graded activity based on work and sports activities on a scale of 0 to 10. Zero represents disability because of knee problems and 10 represents national or international level soccer.

SECONDARY OUTCOMES:
meniscal extrusion on mrı | immediately before the surgery to 12-month post-operative period
  Meniscal extrusion is generally defined as significant (≥3 mm) medial displacement of the meniscus with respect to the central margin of the tibial plateaurecording the preop and postop meniscal extusion
Kellgren Lawrence | immediately before the surgery to 12-month post-operative period
  The Kellgren and Lawrence system is a common method of classifying the severity of osteoarthritis (OA) using five grades
Outer Bridge | immediately before the surgery to 12-month post-operative period
  Outer Bridge classification is a grading system for joint cartilage breakdown.grade: 0 normal-grade 4 - more cartilage damage

CONTACTS AND LOCATIONS:
Overall Officials: AHMET EMRE PAKSOY, Principal Investigator — Ataturk University
Locations (1):
- Atatürk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I will share this data when the work is complete